CLINICAL TRIAL: NCT04949529
Title: Falls: A Marker of Preclinical Alzheimer Disease
Brief Title: Falls: A Marker of Preclinical AD
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susan Stark, Associate Professor of Occupational Therapy, Neurology, and Social Work, Washington University School of Medicine
Other Study IDs: 201807135; R01AG057680-01A1 (NIH)
Record Dates: First submitted 2021-04-09; First posted 2021-07-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Fall; Alzheimer Disease
Keywords: Preclinical Alzheimer Disease; Falls; Functional Mobility; Older Adults
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Whole blood sample
  2. Cerebral spinal fluid (CSF)
  3. Stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This longitudinal cohort study investigates cognitively normal participants with and without preclinical Alzheimer disease (AD) in order to examine: (1) the relationship between falls and functional mobility in preclinical stages of AD; and (2) a hypothesized model of central and peripheral mechanism(s) underlying falls and functional mobility in preclinical stages of AD.

DETAILED DESCRIPTION:
Alzheimer disease (AD) is a slowly progressive neurodegenerative disease. Conversion to symptomatic AD occurs slowly over years through a series of preclinical stages marked by changes in molecular biomarkers. It is unknown whether functional mobility and falls are preclinical markers of AD.

This longitudinal clinical study evaluates a cohort of cognitively normal individuals who are currently undergoing comprehensive clinical, neuropsychological, and biomarker evaluations at the Knight Alzheimer's Disease Research Center (Knight ADRC). They receive an annual in-home evaluation of fall risks and functional mobility and prospective ascertainment of falls. Comparisons of assessments of functional mobility will be performed with regard to measures of brain pathology (i.e., amyloidosis, tau, and neurodegeneration) to allow researchers to characterize when changes in falls and functional mobility occur during preclinical stages of AD.

This study also examines the central and peripheral system mechanism(s) underlying falls and functional mobility in preclinical AD using structural equation modeling.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older
2. cognitively normal (Clinical Dementia Rating [CDR] score of 0)

   * A pilot sub-study collecting stool will also enroll a few individuals with CDR>0 for comparison.
3. have biomarkers (CSF), and/or neuroimaging (positron emission tomography [PET] and/or magnetic resonance imaging [MRI]) within 2 years of enrolling in this study.

Exclusion Criteria:

* History of Parkinson's disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A cohort of cognitively normal community-dwelling older adults who are currently undergoing comprehensive clinical, neuropsychological, and biomarker evaluations at the Knight Alzheimer's Disease Research Center (Knight ADRC) at Washington University in St. Louis.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number and Severity of Falls | Cumulative falls at 4 years post-enrollment
  Prospective monthly fall reporting will be collected using an automated phone/email system. Severity of falls will be calculated using a previously published algorithm.
Change from baseline: Dynamic balance and mobility | 4 years post-enrollment
  Dynamic balance and mobility will be assessed using the Performance Oriented Mobility Assessment (POMA), a task-oriented assessment.
Change from baseline: Gait Speed | 4 years post-enrollment
  Gait speed will be collected using the Timed Up and Go (TUG) test.
Change from baseline: Dual-task gait | 4 years post-enrollment
  Dual-task gait will be collected using the Timed Up and Go Cognitive (TUGcog) and Timed Up and Go Manual (TUGman)

SECONDARY OUTCOMES:
Fall Risk Composite Score | 4 years post-enrollment
  A fall risk composite score will be calculated using established cut-off values, dichotomized as 0 (no risk), or 1 (fall risk), and summed. Higher score indicate higher fall risk. Constructs that will be included are: vision, alcohol abuse, urinary incontinence, depression, pain, medication, functional capacity with activities of daily living, previous falls, home hazards, and self-efficacy.
Change from baseline: Standing balance and vestibular function | 4 years post-enrollment
  Center of pressure path will be measured using Balance Tracking System (BTrackS)
Change from baseline: Lower extremity strength | 4 years post-enrollment
  Lower extremity strength will be assessed using the 30-Second Chair Stand test and minimal change in the peak torque value
Change from baseline: Grip strength | 4 years post-enrollment
  Pounds of force will be measured using a handheld dynamometer
Change from baseline: Vision | 4 years post-enrollment
  Visual acuity will be collected using the Early Treatment Diabetic Retinopathy Study (ETDRS) test, and contrast sensitivity will be measured using the Pelli-Robson test
Change from baseline: Sensation | 4 years post-enrollment
  8-item questionnaire and sensation testing (vibration [feet] and sharp [arms and legs])
Change from baseline: Depression | 4 years post-enrollment
  Frequency of symptoms will be assessed using The Patient Health Questionnaire (PHQ-9) and Geriatric Depression Scale (GDS)
Change in baseline: Functional performance | 4 years post-enrollment
  Independence, safety, and adequacy with shopping, checkbook balancing, and medication management will be assessed using the Performance Assessment of Self-Care Skills (PASS)
Change from baseline: Falls behavior | 4 years post-enrollment
  Behaviors to prevent falls will be measured using the Falls Behavioral Scale for Older People (FaB)
Change from baseline: Olfaction | 2 years post-enrollment
  Olfaction will be assessed using the University of Pennsylvania Smell Identification Test (UPSIT)
Change from baseline: Hearing | 4 years post-enrollment
  Hearing impairment will be assessed using The Hearing Handicap Inventory for the Elderly (HHIE-S)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Stark, PhD, Principal Investigator — Washington University School of Medicine; Beau Ances, MD, PhD, MSc, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bollinger RM, Keleman A, Thompson R, Westerhaus E, Fagan AM, Benzinger TL, Schindler SE, Xiong C, Balota D, Morris JC, Ances BM, Stark SL. Falls: a marker of preclinical Alzheimer disease: a cohort study protocol. BMJ Open. 2021 Sep 15;11(9):e050820. doi: 10.1136/bmjopen-2021-050820. PMID 34526343